CLINICAL TRIAL: NCT04564274
Title: Natural History Study: COV2Base-a Rare Disease by COVID Study
Brief Title: COV2Base-A Rare Disease by COVID Study
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000091; 000091-H
Record Dates: First submitted 2020-09-24; First posted 2020-09-25 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Chronic Health Conditions; Older Age is Associated With Increased Pathogenicity
Keywords: Modifier of Disease; Precision Medicine; Common Diseases; Increase Risk of Severe Outcomes; Gene-Based Risk; Natural History

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: patients with rare and common diseases

SUMMARY:
Background:

SARS-CoV-2 is the virus that causes COVID. It has caused a global pandemic. Most people have no to mild symptoms. But some people need to be hospitalized, and a small number need critical care. Older age as well as some socio-demographic factors and chronic health conditions may play a role in the severity of COVID. In this study, researchers want to assess sociodemographic-, population-, disease-, and gene-based risks for features associated with severe SARS-CoV-2 outcomes. As more is understood about COVID, researchers also want to learn more about people s experiences with COVID vaccines, long-haul symptoms, and other related disease features.

Objective:

To measure the frequency and severity of COVID infection in people with rare and common diseases, looking for conditions that increase risk of severe outcomes. To describe experiences with COVID vaccines, symptoms, and other features of COVID in people with rare and common diseases.

Eligibility:

People greater than 1 month of age, both with and without rare disease, who have access to the Internet.

Design:

This study will take place online.

Participants will visit a website. They will fill out a survey. It should take less than 30 minutes to complete. They will answer questions about their current health and COVID experiences. They will answer questions about their demographic and location features that may impact their exposure to the virus. All questions are optional.

Participants may repeat the survey if their responses indicate a need for follow-up.

Participants medical records may be reviewed.

Participants may be contacted for future studies related to:

COVID

Their underlying health conditions

A new exposure that is being studied....

DETAILED DESCRIPTION:
Study Description:

This protocol will collect information on frequency and severity of COVID infection for patients with rare diseases and community controls.

Study Objectives:

Primary Objective: To quantify the frequency and severity of COVID infection in patients with rare and common diseases, looking for conditions that increase risk of severe outcomes.

Secondary Objective: To identify gene-, tissue- or sociodemographic level features that increase risk of severe COVID outcomes that may inform future genetic modifier studies.

Tertiary Objective (exploratory): To investigate the role of pre- existing disease- or socioeconomic- factors that contribute to COVID- related stress and to evaluate whether individuals with the conditions studied experience more extreme symptoms around the time of COVID vaccine.

Endpoints:

Primary Endpoint: Frequency of severe infection (hospitalization +/- ICU stay and/or COVID-related death) secondary to COVID in patients with a shared disease designation.

Secondary Endpoint: Frequency of severe infection (hospitalization +/- ICU stay and/or COVID-related death) secondary to COVID in patients with shared organ system involvement, secondary comorbidities, or sociodemographic differences.

AND Frequency of any infection or symptoms (including long haul symptoms) secondary to COVID in study patients as grouped by genetic diagnosis, organ system involvement, secondary comorbidities, or sociodemographic features.

Tertiary Endpoints (exploratory): Frequency and degree of COVID related stress based on pre-existing disease-, organ system-, or socioeconomic- factors and frequency of extreme symptoms following one of the COVID vaccines based on pre-existing disease-organ system-, or socioeconomic- factors.

Study Population:

The study will include people greater than 1 month old, with and without rare disease. Some members of the study population have cognitive impairment on the basis of their rare disease.

Description of Sites/Facilities Enrolling Participants:

All consent and study procedures/questionnaire will be performed online.

Study Duration:

The study will enroll for up to 13 months.

Participant Duration:

After consent, participants (or their legal authorized representative) will be asked to fill out an online questionnaire that should take <30 minutes. We may re-send the survey to the participants in 6 - 12 months. Filling out the second round questionnaire is preferred but not required. New enrollees at the time the 2nd questionnaire is sent will fill out the questionnaire once at Time 2. If a signal for increased symptoms is identified in one or more studied groups, individuals from that group may be re-contacted with additional questions or request for medical records within the 13 month window. Participants will be consented for re-contact.

ELIGIBILITY:
* INCLUSION CRITERIA:

The person being reported upon must be 1 month of age or older. The reporter must have access to the internet and be able to read and answer questions in English or Spanish.

EXCLUSION CRITERIA:

Individuals unwilling to allow sharing of their research data should not participate. With the use of online consents for large numbers of individuals, opting in or out of sharing for this low risk study creates a burden for this research study as well as the ability to share data with other related research studies for meta-analysis.

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study groups (those being reported upon) include those with known rare medical conditions and those without (community populations). Some individuals being reported on may be children or those with cognitive impairment.
Sampling Method: Non-Probability Sample
Enrollment: 1748 (Actual)
Dates: Start 2020-10-04 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-05-20 (Actual)

PRIMARY OUTCOMES:
To quantify the frequency and severity of COVID infection in patients with rare and common diseases, looking for conditions that increase risk of severe outcomes. | 12 months
  To quantify the frequency and severity of COVID infection in patients with rare and common diseases, looking for conditions that increase risk of severe outcomes.

SECONDARY OUTCOMES:
To identify gene-, tissue- or sociodemographic level features that increase risk of severe COVID outcomes that may inform future genetic modifier studies. | 13 months
  To identify gene-, tissue- or sociodemographic level features that increase risk of severe COVID outcomes that may inform future genetic modifier studies.

CONTACTS AND LOCATIONS:
Overall Officials: Beth A Kozel, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided